CLINICAL TRIAL: NCT07348367
Title: A Randomized Comparison of Radical Prostatectomy and Precision Prostatectomy in Low- and Intermediate-risk Prostate Cancers.
Brief Title: A Comparison of Radical Prostatectomy and Precision Prostatectomy in Low- and Intermediate-risk Prostate Cancers.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Firas Abdollah, M.D., F.E.B.U. Vice-Chair, Academics and Research, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18404-01
Record Dates: First submitted 2025-09-30; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: Prostatectomy
Keywords: Prostate Cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical Prostatectomy (Active Comparator): This arm is the control arm and consists of the current standard of care. Patients in this arm receive a radical prostatectomy.
  Interventions: Procedure: Radical Prostatectomy
- Precision Prostatectomy (Experimental): This arm is the treatment arm and consists of patients who receive a Precision Prostatectomy.
  Interventions: Procedure: Precision Prostatectomy

INTERVENTIONS:
Procedure: Radical Prostatectomy — In radical prostatectomies, the entire prostate as well as much of the surrounding tissue is removed.
  Other Names: Prostatectomy
  Arms: Radical Prostatectomy
Procedure: Precision Prostatectomy — The surgical approach is very similar to a radical prostatectomy. The difference is that in precision prostatectomy, some of the prostate, including the nerves which might be integral to continence and erectile function are protected and not removed, unlike with traditional radical prostatectomies.
  Arms: Precision Prostatectomy

SUMMARY:
Prostate cancer (PCa) management for low- and intermediate-risk patients often involves radical prostatectomy (RP), which achieves oncologic control but is associated with significant functional impairments, such as erectile dysfunction (50-70%) and urinary incontinence (5-20%). To address these issues, precision prostatectomy (PP) has emerged as a novel surgical approach that preserves functional structures while removing >90% of prostate tissue.

PP is thought to provide superior functional outcomes with acceptable oncological control by preserving the capsule, seminal vesicle (SV), and the surrounding neuronal nitric oxide synthase (nNOS) producing nerves on the side opposite to the dominant nodule while maximizing prostatic tissue removal. Early reports of PP demonstrate promising functional outcomes, with 90% of patients retaining sexual potency (Sexual Health Inventory for Men [SHIM] score ≥17) and 100% achieving continence (0-1 pads/day) by 12 months postoperatively. Importantly, PP only requires a different surgical technique, no more equipment, time, or labor is required. This means that there is no additional charge to patients, and it is covered the same by health insurance.

While there are early results suggesting the superiority of PP, no randomized trials have yet to be performed. This study has two main aims: to demonstrate superiority of PP in terms of functional recovery while also establishing non-inferiority in oncologic outcomes compared to RP. This dual objective reflects the potential of PP to improve quality of life without compromising cancer control.

Eligible patients will be randomized to either RP, which is the current standard of care, or PP using random blocked randomization using the Zelen design.

The outcomes of interest will be measured at 12 months post-surgery. Functional outcomes will be measured using SHIM scores at 12 months and the number of pads used per day. Meanwhile, oncological outcomes will be measured by whether patients have received secondary prostate cancer treatment at 12 months post-surgery. These items are collected as part of standard of care of all patients 12 months after prostatectomy. RP and PP patients' sexual function recovery (SHIM ≥17 vs SHIM < 17), as well as the proportion reaching continence (≤1 pad per day, > 1 pad per day) will be compared.

RP has been shown to be effective in terms of oncological outcomes, though it has also been shown to be related to incontinence and erectile dysfunction. Early results have suggested that PP is superior in terms of functional outcomes while being as good as RP in terms of oncological outcomes, though no randomized trials have been conducted. This trial will address this literature gap and could lead to patients receiving care that is as effective ontologically and superior in terms of functional recovery as the current standard of care. This could lead to improved quality of life for patients after surgery. Considering that prostate cancer is the most common non-cutaneous carcinoma among men in the United States, this has the potential to help thousands of men per year by improving their quality of life without sacrificing oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients receiving treatment at Henry Ford Health from the investigator or co-investigator who opt for surgery.
* Prostate-specific antigen (PSA) ≤20 ng/mL
* Clinical stage ≤cT2
* Dominant unilateral lesion with Gleason ≤4+3 on biopsy
* No Gleason ≥4 contralaterally
* Preoperative SHIM score ≥17 (with or without phosphodiesterase-5 inhibitor use)

Exclusion Criteria:

* • Androgen deprivation therapy within 6 months.

  * Nodal positive disease
  * Metastatic disease
  * Prior prostate cancer therapy (e.g., radiation, HIFU).
  * Significant comorbidities precluding surgery or life expectancy <5 years as defined by the Prostate Cancer Comorbidity Index [5].
  * Any previous cancer diagnosis.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sexual Health | Before surgery, 3 months post-surgery, 12 months post-surgery
  Patients' sexual health and function is measured by the Sexual Health Inventory for Men (SHIM). A SHIM score > 16 is considered sexually healthy.
Social Continence | 12 months post-surgery.
  Continence is determined by the number of pads used per day by patients. Social continence is defined as < 2 pads per day.

SECONDARY OUTCOMES:
Oncological outcomes | 12-months post-surgery
  The number of patients who undergo secondary treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
At this time we do not plan on making a deidentified dataset and PHI cannot be shared per institutional policies. We will consider sharing deidentified data upon request.

REFERENCES:
- [Background] Sood A, Jeong W, Keeley J, Abdollah F, Hassan O, Gupta N, Menon M. Subtotal surgical therapy for localized prostate cancer: a single-center precision prostatectomy experience in 25 patients, and SEER-registry data analysis. Transl Androl Urol. 2021 Jul;10(7):3155-3166. doi: 10.21037/tau-20-1476. PMID 34430418
- [Background] Capogrosso P, Vertosick EA, Benfante NE, Eastham JA, Scardino PJ, Vickers AJ, Mulhall JP. Are We Improving Erectile Function Recovery After Radical Prostatectomy? Analysis of Patients Treated over the Last Decade. Eur Urol. 2019 Feb;75(2):221-228. doi: 10.1016/j.eururo.2018.08.039. Epub 2018 Sep 17. PMID 30237021
- [Background] Resnick MJ, Koyama T, Fan KH, Albertsen PC, Goodman M, Hamilton AS, Hoffman RM, Potosky AL, Stanford JL, Stroup AM, Van Horn RL, Penson DF. Long-term functional outcomes after treatment for localized prostate cancer. N Engl J Med. 2013 Jan 31;368(5):436-45. doi: 10.1056/NEJMoa1209978. PMID 23363497
- [Background] Menon M, Shrivastava A, Tewari A, Sarle R, Hemal A, Peabody JO, Vallancien G. Laparoscopic and robot assisted radical prostatectomy: establishment of a structured program and preliminary analysis of outcomes. J Urol. 2002 Sep;168(3):945-9. doi: 10.1016/S0022-5347(05)64548-X. PMID 12187196
- [Background] Xiao H, Tan F, Goovaerts P, Ali A, Adunlin G, Huang Y, Gwede C. Construction of a comorbidity index for prostate cancer patients linking state cancer registry with inpatient and outpatient data. J Registry Manag. 2013 Winter;40(4):159-64. PMID 24625768
- [Background] Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Pena BM. Development and evaluation of an abridged, 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res. 1999 Dec;11(6):319-26. doi: 10.1038/sj.ijir.3900472. PMID 10637462
- [Background] Sood A, Jeong W, Taneja K, Abdollah F, Palma-Zamora I, Arora S, Gupta N, Menon M. The Precision Prostatectomy: an IDEAL Stage 0, 1 and 2a Study. BMJ Surg Interv Health Technol. 2019 Aug 19;1(1):e000002. doi: 10.1136/bmjsit-2019-000002. eCollection 2019. PMID 35047770